CLINICAL TRIAL: NCT03048656
Title: Does the Structural Leg-length Discrepancy Affect the Postural Control? Preliminary Study
Brief Title: The Postural Control in Individuals With the Structural Leg-length Discrepancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Małgorzata Eliks, Assistant, MSc, Poznan University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 418/14
Record Dates: First submitted 2017-02-06; First posted 2017-02-09 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Leg Length Inequality
MeSH Terms: conditions — Leg Length Inequality

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individuals with leg-length discrepancy (Experimental): Patients of Department of Paediatric Orthopaedics and Traumatology, Poznan University of Medical Sciences diagnosed with leg-length discrepancy. The examination of participants included a measurement of the length of lower limbs and the weight distribution as well as performing the static posturography.
  Interventions: Other: static posturography
- control group (Active Comparator): The group with healthy individuals; without leg-length discrepancy. The examination of participants included a measurement of the weight distribution as well as performing the static posturography.
  Interventions: Other: static posturography

INTERVENTIONS:
Other: static posturography — The measurement of the weight distribution and the static posturography was performed on the balance platform Good Balance by Metitur . The device is comprised of the triangular force platform with electronic system and computer software. The body weight distribution was evaluated in the upright standing with eyes open, feet placed 20 cm from each other.The individual stood motionlessly for 15 s, then the measurement was recorded. The static posturography was performed with 3 various positions of feet, both with eyes open and eyes closed. (1) Position : normal standing - an upright standing with feet placed parallel 20 cm apart for 30 s. (2) Position: tandem - a stance with one foot placed ahead of the other. for 20 s. (3) Position: one leg standing: stance on the one leg for 20 s.

SUMMARY:
The structural leg-length inequality caused by the shortening of a segment of an extremity, results in an altered position of lower limb joints, the pelvis and the spine in static as well as dynamic conditions. That may induce a disturbance of the postural control.

The objective of this study is to investigate the effect of the structural LLD on the control of the posture.

DETAILED DESCRIPTION:
The measurement of the weight distribution and the static posturography is performed on the balance platform Good Balance by Metitur . The device is comprised of the triangular force platform (800 mm x 800 mm x 800 mm) with electronic system and computer software. The body weight distribution is evaluated in the upright standing with eyes open, feet placed 20 cm from each other or narrower in children, with upper extremities in relaxed position by sides. The individual stands motionlessly for 15 s, then the measurement is recorded. The results of each lower extremity loading and a difference in weight bearing between extremities are expressed in percentages (%) .

The static posturography examination is performed with 3 various positions of feet, both with eyes open (EO) and eyes closed (EC). (1) Position : normal standing - an upright standing with feet placed parallel 20 cm apart. (2) Position: tandem - a stance with one foot placed ahead of the other, medial edge of feet was put on the midline of the balance platform. In the experimental group 2 trials were recorded: (a) foot of the shorter leg in the front, (b) foot of the shorter leg in the rear. In the control group also 2 trials are performed: (c) foot of the right leg in the front, (d) foot of the left leg in the front. (3) Position: one leg standing: stance on the one leg, foot placed 10 cm from midline of the platform, the other - 90 degrees flexion of the knee and the hip, test performed only with EO. Every participant is supposed to stand motionlessly for 30 s in normal standing , or for 20 s in tandem .and one leg standing position. Conditions of the posturographic examination involved : quiet and normally lit room , standing barefoot , the eyesight directed at a point in the distance of 2 m , glasses or contact lenses are worn if they are normally needed, arms held in the front of the body with hands together in order to limit movements of upper extremities . The recording is initiated when a stable position is attained . Each test is performed once .

Mean velocity (mm/s) of COP sway is measured as a quantitative parameter of the postural control assessment . Mean COP sway velocity is recorded both in anteroposterior (AP) and mediolateral (ML) directions .

ELIGIBILITY:
Inclusion Criteria:

* for patients: structural leg length discrepancy
* for healthy volunteers: symmetrical length of lower limbs

Exclusion Criteria:

* for patients: achondroplasia, non-union, idiopathic scoliosis, extremity shortening in the course of neurological disease (e.g. Cerebral Palsy), vestibular disorder (e.g. Ménière's disease), diabetes, sensory disorder, intake of medications affecting psychomotor activity, dizziness, neurological diseases (e.g. epilepsy), BMI>30, using mobility aids (e.g. crutches)
* for healthy volunteers: leg-length discrepancy, scoliosis, faulty posture, vestibular disorders, diabetes, intake of medications affecting psychomotor activity, dizziness, sensory disorders, neurological disease, BMI>30.

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2017-01-25 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of mean COP velocity in anteroposterior and mediolateral directions during stance in subjects | 1.02.2017
  Mean COP velocity [mm/s] is recorded in anteroposterior (AP) and mediolateral (ML) directions within posturographic evaluation in examination of every participant.

SECONDARY OUTCOMES:
Evaluation of weight distribution during stance in subjects | 1.02.2017
  The weight loading of each limb is assessed in every participants. The result is expressed in kilograms [kg].

CONTACTS AND LOCATIONS:
Overall Officials: Przemysław Lisiński, PhD, Study Director — Poznan University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahar RK, Kirby RL, MacLeod DA. Simulated leg-length discrepancy: its effect on mean center-of-pressure position and postural sway. Arch Phys Med Rehabil. 1985 Dec;66(12):822-4. PMID 4074116
- [Background] Murrell P, Cornwall MW, Doucet SK. Leg-length discrepancy: effect on the amplitude of postural sway. Arch Phys Med Rehabil. 1991 Aug;72(9):646-8. PMID 1859258
- [Background] Sabharwal S, Kumar A. Methods for assessing leg length discrepancy. Clin Orthop Relat Res. 2008 Dec;466(12):2910-22. doi: 10.1007/s11999-008-0524-9. Epub 2008 Oct 4. PMID 18836788
- [Background] Lisinski P, Huber J, Gajewska E, Szlapinski P. The body balance training effect on improvement of motor functions in paretic extremities in patients after stroke. A randomized, single blinded trial. Clin Neurol Neurosurg. 2012 Jan;114(1):31-6. doi: 10.1016/j.clineuro.2011.09.002. Epub 2011 Oct 2. PMID 21963145
- [Background] Swaminathan V, Cartwright-Terry M, Moorehead JD, Bowey A, Scott SJ. The effect of leg length discrepancy upon load distribution in the static phase (standing). Gait Posture. 2014 Sep;40(4):561-3. doi: 10.1016/j.gaitpost.2014.06.020. Epub 2014 Jul 17. PMID 25082323
- [Background] Pajala S, Era P, Koskenvuo M, Kaprio J, Tolvanen A, Heikkinen E, Tiainen K, Rantanen T. Contribution of genetic and environmental effects to postural balance in older female twins. J Appl Physiol (1985). 2004 Jan;96(1):308-15. doi: 10.1152/japplphysiol.00660.2003. Epub 2003 Sep 5. PMID 12959956
- [Background] Betsch M, Rapp W, Przibylla A, Jungbluth P, Hakimi M, Schneppendahl J, Thelen S, Wild M. Determination of the amount of leg length inequality that alters spinal posture in healthy subjects using rasterstereography. Eur Spine J. 2013 Jun;22(6):1354-61. doi: 10.1007/s00586-013-2720-x. Epub 2013 Mar 13. PMID 23479027
- [Background] Betsch M, Wild M, Grosse B, Rapp W, Horstmann T. The effect of simulating leg length inequality on spinal posture and pelvic position: a dynamic rasterstereographic analysis. Eur Spine J. 2012 Apr;21(4):691-7. doi: 10.1007/s00586-011-1912-5. Epub 2011 Jul 17. PMID 21769443
- [Background] Young RS, Andrew PD, Cummings GS. Effect of simulating leg length inequality on pelvic torsion and trunk mobility. Gait Posture. 2000 Jun;11(3):217-23. doi: 10.1016/s0966-6362(00)00048-5. PMID 10802434
- [Derived] Eliks M, Ostiak-Tomaszewska W, Lisinski P, Koczewski P. Does structural leg-length discrepancy affect postural control? Preliminary study. BMC Musculoskelet Disord. 2017 Aug 9;18(1):346. doi: 10.1186/s12891-017-1707-x. PMID 28793888